CLINICAL TRIAL: NCT03421340
Title: Prospective, Multi-center, Randomized Controlled Study Comparing Endoscopic Clearance of Non-Complex Biliary Stones Using Fluoroscopy/Radiation-Free Direct Solitary Cholangioscopy (DSC) to Standard of Care Endoscopic Retrograde Cholangiography (ERC)
Brief Title: Non-Complex Biliary Stones DSC vs ERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E7131
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-09

CONDITIONS: Biliary Stones
Keywords: ERCP; DSC; Spy Glass; Biliary Stones; Choledocholithiasis; Non-Complex; Stones
MeSH Terms: conditions — Cholecystolithiasis; Choledocholithiasis; Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ERC Arm (Other): After screening examination and confirmed presence of non-complex bile duct stone by image, patients will be randomly assigned by stratified randomization to Endoscopic Retrograde Cholangioscopy (ERC) treatment.
  Interventions: Device: ERC
- DSC Arm (Other): After screening examination and confirmed presence of non-complex bile duct stone by imagine, patients will be randomly assigned by stratified randomization to fluoroscopy/radiation-free direct solitary cholangioscopy (DSC).
  Interventions: Device: DSC

INTERVENTIONS:
Device: DSC — Stone removal without fluoroscopy using the SpyGlass device.
  Other Names: Direct Solitary Cholangioscopy
  Arms: DSC Arm
Device: ERC — Standard of care stone removal with fluoroscopy.
  Other Names: Endoscopic Retrograde Cholangiography
  Arms: ERC Arm

SUMMARY:
To prospectively compare non-complex biliary stone clearance using fluoroscopy/radiation-free direct solitary cholangioscopy (DSC) utilizing the SpyGlass™ system with non-complex biliary stone clearance using standard endoscopic retrograde cholangiography (ERC).

DETAILED DESCRIPTION:
The objective of this study is to prospectively compare non-complex biliary stone clearance using fluoroscopy/radiation-free direct solitary cholangioscopy (DSC) utilizing the SpyGlass™ system with non-complex biliary stone clearance using standard endoscopic retrograde cholangioscopy (ERC).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Abdominal pain consistent with choledocholithiasis (procedure possible within 72 hours of onset of symptoms and imaging suggesting choledocholithiasis, contingent on persistent abdominal pain)
3. Abnormal LFTs
4. Non-complex biliary stone disease, defined as 5 or fewer stones in the common bile or common hepatic duct with largest stone no larger than 10 mm in size. If stones not seen on imaging (US, CT) the bile duct diameter should be ≤12 mm*

   * Given the poor sensitivity (approximately 20%) for biliary stones of CT and US, the diameter of the dilated CBD is used as a surrogate for largest stone diameter
5. Availability of non-invasive imaging to determine the diameter of the bile duct and number and size of bile duct stones if visible on imaging

   1. If probability of stones is high per investigator assessment based on ASGE criteria, any standard of practice imaging modality (eg. abdominal US) is acceptable.
   2. If the probability of stones is either intermediate or low per investigator assessment based on ASGE criteria, MRCP or EUS imaging is required to confirm presence of stones.
6. Willing and able to comply with the study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

1. Potentially vulnerable subjects, including but not limited to pregnant women and subjects in whom an endoscopic procedure is contraindicated
2. Location of the stones in intrahepatic ducts, cystic duct or proximal to strictures
3. Bile duct stricture noted distal to stone on MRCP, which would make extraction without lithotripsy impossible
4. Ongoing cholangitis at time of randomization, manifested by fever with tachycardia and hypotension or evidence of pus at the ampulla
5. Patients with prior biliary sphincterotomy
6. Patients with Primary Sclerosing Cholangitis (PSC)
7. Acute pancreatitis, defined as abdominal pain and serum concentration of pancreatic enzymes [lipase (required), amylase (optional)] three or more times the upper limit of normal
8. Surgically altered gastro-duodenal luminal anatomy other than prior Billroth I reconstruction, as these would be anticipated to lead to more complicated procedures
9. Coagulopathy or ongoing need for anti-coagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Principal Investigator — Stanford University; Nirav Thosani, MD, Principal Investigator — Univeristy of Texas Health Sciences; Raj J Shah, MD, Principal Investigator — University of Colorado, Denver; Mohan Ramchandani, MD, Principal Investigator — Asian Institure of Gastroenterology; Guido Costamagna, MD, Principal Investigator — Fundazione Policlinico Universitario; Rungsun Rerknimitr, MD, Principal Investigator — King Chulalongkorn Memorial Hospital; Janak N Shah, MD, Principal Investigator — Ochsner Health System; Mahesh Goenka, MD, Principal Investigator — Apollo Gleneagles Hospitals, Kolkata
Locations (8):
- United States (4):
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital, Denver, Aurora, Colorado
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Ertan Digestive Disease Center - University of Texas Health Science Center, Houston, Texas
- India (2):
  - Asian Institute of Gastroenterology, Hyderabad, Somajiguda
  - Apollo Gleneagles Hospitals Kolkata, Kolkata, West Bengal
- Fundazione Policlinico Universitario Agostino Gemelli, Rome, Italy
- King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Derived] Banerjee S, Goenka MK, Ramchandani M, Shah RJ, Lakhtakia S, Ridtitid W, Shah JN, Thosani N, Wagh MS, Costamagna G, Peetermans JA, Rousseau MJ, Rerknimitr R. Fluoroscopy-free Direct Solitary Cholangioscopy versus Endoscopic Retrograde Cholangiography for Clearance of Noncomplex Biliary Stones: A Noninferiority Randomized Controlled Trial. Gastrointest Endosc. 2026 Jan 16:S0016-5107(25)02534-9. doi: 10.1016/j.gie.2025.12.283. Online ahead of print. PMID 41548725
- [Derived] Ridtitid W, Rerknimitr R, Ramchandani M, Lakhtakia S, Shah RJ, Shah JN, Thosani N, Goenka MK, Costamagna G, Wagh MS, Perri V, Peetermans J, Goswamy PG, Liu Z, Yin S, Banerjee S. Endoscopic clearance of non-complex biliary stones using fluoroscopy-free direct solitary cholangioscopy: Initial multicenter experience. DEN Open. 2023 Jun 1;4(1):e241. doi: 10.1002/deo2.241. eCollection 2024 Apr. PMID 37273518

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ERC Arm | DSC Arm
Started | 126 | 124
Completed | 115 | 117
Not Completed | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ERC Arm | DSC Arm | Total
Number analyzed (Participants) | 126 | 124 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (16.7) | 50.3 (18) | 52 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 79 | 150
  Male | 55 | 45 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40 | 39 | 79
  Italy | 0 | 1 | 1
  Thailand | 27 | 26 | 53
  India | 59 | 58 | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Stone Clearance
Description: Prospectively compare DSC vs. ERC
Time Frame: 30 Days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | ERC Arm | DSC Arm
Number analyzed (Participants) | 126 | 124
Participants | 112 | 108
Statistical Analysis 1: Comparison: ERC Arm vs DSC Arm; Test type: Non-Inferiority — Non-Inferiority Margin of 10%; p = 0.029, exact; Risk Difference (RD) = 1.8

2. Secondary Outcome: Rate of Serious Adverse Events
Description: To evaluate all SAEs including death, severity, onset, time to resolution.
Time Frame: 30 Days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | ERC Arm | DSC Arm
Number analyzed (Participants) | 126 | 124
Participants | 5 | 7
Statistical Analysis 1: Comparison: ERC Arm vs DSC Arm; Test type: Superiority — Not powered; Risk Difference (RD) = -1.7, 95% CI 2-sided [-8 to 4.1]

3. Secondary Outcome: Radiation Exposure
Description: Total Fluoroscopy time
Time Frame: 3 hours
Measure: Median (Full Range); unit: seconds
Arm/Group | ERC Arm | DSC Arm
Number analyzed (Participants) | 126 | 124
seconds | 133 [0 to 720] | 0 [0 to 454]
Statistical Analysis 1: Comparison: ERC Arm vs DSC Arm; Test type: Superiority; Median Difference (Net) = 133, 95% CI 2-sided [120 to 143]

4. Secondary Outcome: Duration of Procedure
Description: Defined as time from duodenoscope in to completion of stone clearance.
Time Frame: 3 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | ERC Arm | DSC Arm
Number analyzed (Participants) | 126 | 124
minutes | 11.9 [3.8 to 137.9] | 22.1 [6.0 to 67.0]
Statistical Analysis 1: Comparison: ERC Arm vs DSC Arm; Test type: Superiority; Median Difference (Final Values) = -10.2, 95% CI 2-sided [-11.6 to -7.5]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | ERC Arm | DSC Arm
All-Cause Mortality (participants affected / at risk) | 1/126 | 1/124
Serious Adverse Events (participants affected / at risk) | 5/126 | 7/124
Other Adverse Events (participants affected / at risk) | 0/126 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERC Arm (N=126) | DSC Arm (N=124)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 5 (5)
Duodenal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03421340/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03421340/SAP_002.pdf